CLINICAL TRIAL: NCT02191813
Title: The Ability of Seresis to Act as a Skin Protection Agent: a Double-blind, Parallel Group, Placebo-controlled Trial in Healthy, Young Female Volunteers
Brief Title: Study to Determine the Ability of Seresis to Act as a Skin Protection Agent in Healthy Young Female Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1135.3
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Seresis® (Experimental)
  Interventions: Drug: Seresis®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seresis®
  Arms: Seresis®
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to detect the efficacy of Seresis® in reducing the damage produced on the skin by Matrix-metalloproteinases (MMP) and by oxidative stress (marker: heme oxygenase-1 expression) activated by UV radiation

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers between 18 and 30 years
* With skin type I or skin type II
* Body Mass Index > 25
* Non-smokers
* Volunteers who have given their written informed consent according to Good Clinical Practice (GCP) and local regulations

Exclusion Criteria:

* Any serious disorder that may interfere with her participation to the trial and evaluation of the safety of the test drug (e.g. liver and/or renal disease, hypervitaminosis A, psychic disorder, etc.), and/or treatment with chronic medication
* Pre-treatment (less than 2 weeks prior to inclusion in this trial) and/or concomitant treatment with any drug that may influence the trial symptomatology and may interfere with evaluation of the safety of the test drug (e.g. vitamins and minerals supplementation)
* Relevant allergy or known hypersensitivity to the investigational drug or its excipients
* High performance sports people
* Alcohol and drug abuse according to Diagnostic and Statistics Manual (DSM-IV)
* Female volunteers in child-bearing age not using adequate means of birth control (contraceptive pills, intrauterine device (IUDs), sterilization)
* Pregnancy and/or lactation
* Known abnormal values of the lab tests (if detected after enrolment, subjects will continue the treatment provided there are no medical objections)
* Abnormal values of Aspartate Transferase (SGOT/ASAT), Alanine Transferase (SGPT/ALAT)-, Gamma-glutamyl transpeptidase, Low density Lipoproteins/Triglycerides (LDL/TGL) levels in blood
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial
* Specific dietary requirements that do not allow the volunteers to meet the dietary guidelines set out for this study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2000-03; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Absolute changes in MMP-1 levels (activity and protein expression) measured in skin samples | Day 84
Absolute changes in MMP-9 levels (activity and protein expression) measured in skin samples | Day 84

SECONDARY OUTCOMES:
Changes in MMP-1 levels measured in skin samples | up to day 84
Changes in MMP-9 levels measured in skin samples | up to day 84
Changes in MMP-3 levels measured in skin samples | up to day 84
Changes in pro-MMPs levels measured in skin samples | up to day 84
Changes in tissue inhibitor (TIMP-1) levels measured in skin samples | up to day 84
Heme oxygenase-1 level measured in skin samples | up to day 84
Density of Langerhans cells measured in skin samples | up to day 84
Cell proliferation and differentiation measured in skin samples | up to day 84
Plasma levels of vitamin E | up to day 84
Plasma levels of beta-carotene | up to day 84
Number of subjects with adverse events | up to 112 days
Number of subjects with abnormal changes in laboratory parameters | up to day 98
Assessment of tolerability by investigator on a 4-point scale | Day 84
Assessment of tolerability by volunteer on a 4-point scale | Day 84
Recall antigene (skin immune status) measured in the skin sample | up to 84 days
Assessment of light sensitivity | up to 84 days